CLINICAL TRIAL: NCT04010526
Title: Double-blind Randomised Placebo Controlled Study Evaluating Local Co-administration of Autologous ADIpose Derived Stromal Vascular Fraction With Microfat for Refractory Perianal CROHN's Fistulas.
Brief Title: Evaluation of Local Co-administration of Autologous ADIpose Derived Stromal Vascular Fraction With Microfat for Refractory Perianal CROHN's Fistulas.
Acronym: ADICROHN2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RCAPHM18_0013
Record Dates: First submitted 2018-09-06; First posted 2019-07-08 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): CD patients with complex refractory perianal fistula refractory to conventional medical and surgical therapy referred to the gastroenterology departments of the 3 centers in charge of treatment local co-administration of autologous ADIpose will be performed
  Interventions: Combination Product: local co-administration of autologous ADIpose
- placebo (Placebo Comparator): CD patients with complex refractory perianal fistula refractory to conventional medical and surgical therapy referred to the gastroenterology departments of the 3 centers in charge of treatment local co-administration of placebo will be performed
  Interventions: Other: placebo

INTERVENTIONS:
Combination Product: local co-administration of autologous ADIpose — local co-administration of autologous ADIpose derived stromal vascular fraction and microfat for refractory perianal CROHN's fistulas Each batch of the final product is composed of one 5 mL syringes containing 25,9 +/- 10,7 millions viable cells. Each syringe will be obstructed with a sterile stopper and packaged in an external packaging.
  Arms: treatment
Other: placebo — local co-administration of placebo The study placebo will consist of a saline solution for intralesional administration and will follow the same administration schema described for the SFV
  Arms: placebo

SUMMARY:
Autologous ADSVF constitutes an innovative therapeutic strategy that concentrates various types of regenerative stem cells and paracrine factors able to promote angiogenesis and tissue repair. Together with the ease of collection from a minimally manipulated lipoaspirate, the unique properties of ADSVF offer new opportunities for fistulas' healing in patients with CD. The use of ADSVF is currently developed in many clinical fields based on safety and efficacy data.

Our ADICROHN pilot study evaluating safety and tolerance of local administration of autologous ADSVF with microfat in CD patients with complex perianal fistula refractory to conventional medical and surgical therapy showed that this novel therapeutic approach appears feasible and safe.

However the therapeutic potential of local this combined treatment in healing refractory perianal Crohn's fistulas still remains to be demonstrated.

The main objective of this study is to assess the efficacy of local injection of autologous ADSVF and microfat versus placebo for the treatment of complex refractory perianal Crohn's fistulas at week 24.

The efficacy will be assessed on clinical assessment of closure of all the external openings that were drained at baseline, and MRI confirmation of absence of collections > 2 cm of the treated perianal fistulas at week 24.

DETAILED DESCRIPTION:
Autologous ADSVF constitutes an innovative therapeutic strategy that concentrates various types of regenerative stem cells and paracrine factors able to promote angiogenesis and tissue repair. Together with the ease of collection from a minimally manipulated lipoaspirate, the unique properties of ADSVF offer new opportunities for fistulas' healing in patients with CD. The use of ADSVF is currently developed in many clinical fields based on safety and efficacy data.

Our ADICROHN pilot study evaluating safety and tolerance of local administration of autologous ADSVF with microfat in CD patients with complex perianal fistula refractory to conventional medical and surgical therapy showed that this novel therapeutic approach appears feasible and safe.

However the therapeutic potential of local this combined treatment in healing refractory perianal Crohn's fistulas still remains to be demonstrated.

B. Primary objective/endpoint The main objective of this study is to assess the efficacy of local injection of autologous ADSVF and microfat versus placebo for the treatment of complex refractory perianal Crohn's fistulas at week 24 (W24), The efficacy will be assessed on clinical assessment of closure (despite gentle finger compression) of all the external openings that were drained at baseline, and MRI confirmation of absence of collections > 2 cm of the treated perianal fistulas at week 24.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients with Crohn's Disease (CD) diagnosed at least 6 months earlier in accordance with accepted clinical, endoscopic, histological and/or radiologic criteria
* Presence of refractory complex perianal fistulas assessed by clinical assessment during examination under anaesthesia (preparation treatment) and MRI.
* Non-active or mildly active luminal CD defined by a CDAI ≤ 220
* Patients of either sex aged 18 years or older
* Good general state of health according to clinical history and a physical examination
* For women of a childbearing age, they must have negative serum or urine pregnancy test (sensitive to 25 IU human chorionic gonadotropin [hCG]). Both men and women should use appropriate birth control methods defined by the investigator.

Exclusion Criteria:

* Presence of dominant luminal active Crohn's disease requiring immediate therapy
* CDAI > 220
* Patient naïve to specific treatment for perianal fistulising Crohn's disease
* Presence of an abscess or collections > 2 cm, unless resolved in the preparation procedure
* Rectal and/or anal stenosis if this means a limitation for any surgical procedure
* Patient with ongoing steroid treatment or treated with steroids in the last 4 weeks
* Malignant tumour or patients with a prior history of any malignant tumour, including any type of fistula carcinoma
* Current or recent history of abnormal, severe, progressive, uncontrolled infectious, hepatic, haematological, gastrointestinal (except CD), endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral disease
* Congenital or acquired immunodeficiencies
* Contraindication to local anaesthetics or gadolinium (MRI contrast)
* Contraindication to MRI scan, (e.g., due to the presence of pacemakers, hip replacements or severe claustrophobia)
* Pregnant or breastfeeding women
* Contraindication to the anaesthetic or surgical procedure
* BMI < 18 to insure adequate abdominal or other subcutaneous adipose tissue accessible by lipoharvest
* Any active viral infection follows: HIV, HTLV I et II, VHB, VHC and Syphillis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
clinically evaluated | 24 weeks (w)
  number of fistula closure
Magnetic resonance imaging (MRI) | weeks 24
  confirmation of absence of collections > 2 cm of the treated perianal fistulas
Magnetic resonance imaging (MRI) | weeks 52
  confirmation of absence of collections > 2 cm of the treated perianal fistulas

SECONDARY OUTCOMES:
a complete cessation of suppuration | weeks4, weeks12, weeks24, weeks52
closure of all the external openings | weeks4, weeks12
Index PDAI (Perianal Disease Activity ) | weeks4, weeks12, weeks24 and weeks52
improvement of Quality of Life Short Inflammatory Bowel Disease Questionnaire (SIBDQ) (QoL) | weeks4, weeks12, weeks24 and weeks52
Crohn's Disease Activity Index (CDAI) | weeks4, weeks12, weeks24 and weeks52
Reduction of anal incontinence severity (Wexner score) | weeks4, weeks12, weeks24 and weeks52

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France

REFERENCES:
- [Derived] Guillo L, Grimaud F, Houser F, Prost C, Jouve E, Philandrianos C, Abellan M, Veran J, Visee C, Beyer-Berjot L, Desjeux A, Dignat-George F, Leone M, Grimaud JC, Sabatier F, Serrero M, Magalon J. Three-year outcome of local injection of autologous stromal vascular fraction cells and microfat in refractory perianal fistulas of Crohn's disease. Stem Cell Res Ther. 2022 Feb 9;13(1):67. doi: 10.1186/s13287-022-02738-x. PMID 35139888